CLINICAL TRIAL: NCT06993493
Title: An Exploratory Clinical Study to Evaluate the Safety and Efficacy of Autologous CD19 CAR - T in the Treatment of Relapsed/Refractory Autoimmune Diseases
Brief Title: Autologous CD19CAR-T Therapy for Recurrent/Refractory Autoimmune Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Boren Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BRYY-IIT-LCYJ-2024-020
Record Dates: First submitted 2025-02-18; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2024-08

CONDITIONS: Autoimmune Disease
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CD19 CART (Experimental)
  Interventions: Genetic: CD19 CART

INTERVENTIONS:
Genetic: CD19 CART — The dose escalation is carried out according to the principle of "3+3" escalation, with a total of 3 dose groups set up.
  Expected sample size (± 30%, CAR+T cells/kg)
  1. 0.5 × 106 0.4 × 106~0.6 × 106 3-6 cases
  2. 1.0 × 106 0.7 × 106~1.3 × 106 3-6 cases
  3. 2.0 × 106 1.4 × 106~2.6 × 106 3-6 cases The enrollment starts from dose group 1, and if no DLT occurs in the 3 subjects included, they will be transferred to the next dose group. If one of the three subjects in a certain dose group develops DLT, three additional subjects will be added to the group for cell infusion at the same dose. If there is ≥ 1 case of DLT in the 3 additional cases (i.e. ≥ 2/6 cases in this dose group), it will be reduced to the previous dose group. If there are only 3 subjects in the previous dose group at this time, an additional 3 subjects need to be added for the trial; If there are already 6 subjects in the previous dose group, the trial ends and this dose is MTD.

SUMMARY:
This study is a single center, open label exploratory clinical trial aimed at evaluating the safety and efficacy of autologous CD19 CAR-T therapy in subjects with autoimmune diseases.

The study will adopt the traditional dose escalation model "3+3" design, with three dose groups set up, starting at a dose of 0.5 × 106 CAR+T cells/kg, to observe DLT, and conduct a 24 month safety and efficacy follow-up after cell infusion to observe the safety of autologous CD19 CAR-T and conduct preliminary efficacy evaluation.

Three dose groups were set up, with dose group 1 as the starting dose, following the traditional 3+3 design rule for a single intravenous infusion:

Dose group dosage unit (CAR+T cells/kg) Acceptable dose range Expected sample size (± 30%, CAR+T cells/kg)

1. 0.5 × 106 0.4 × 106~0.6 × 106 3-6 cases
2. 1.0 × 106 0.7 × 106~1.3 × 106 3-6 cases
3. 2.0 × 106 1.4 × 106~2.6 × 106 3-6 cases Dose escalation rule The enrollment starts from dose group 1, and if no DLT occurs in the 3 subjects included, they will be transferred to the next dose group. If one of the three subjects in a certain dose group develops DLT, three additional subjects will be added to the group for cell infusion at the same dose. If there is ≥ 1 case of DLT in the 3 additional cases, it will be reduced to the previous dose group. If there are only 3 subjects in the previous dose group at this time, an additional 3 subjects need to be added for the trial; If there are already 6 subjects in the previous dose group, the trial ends and this dose is the maximum tolerated dose (MTD).

Dose escalation is not allowed for the same subject. For safety reasons, the last subject in the previous dose group was observed for at least 28 days after autologous CD19 CAR-T infusion without DLT. The Safety Review Committee (SRC) held a meeting to decide whether to increase to the next dose group.

During the dose escalation phase, SRC determines whether to continue increasing the dose or explore more subjects in a previously explored dose group based on the safety, efficacy, and pharmacokinetic (PK) results obtained for each dose group, and determines the recommended dose (RD) for subsequent studies.

ELIGIBILITY:
Inclusion Criteria:

* Age range of 18 to 65 years old (including 18 and 65 years old), gender is not limited;
* Special criteria for different indications:
* Subjects with relapsed/refractory moderate to severe SLE must meet the following criteria:
* According to the 2019 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) SLE classification criteria, the diagnosis is SLE;
* Positive for anti nuclear antibody (ANA) (titer ≥ 1:80), and/or positive for anti dsDNA antibody, and/or positive for anti Sm antibody during screening;
* The definition of moderate to severe activity is: SLEDAI-2000 score ≥ 8 during screening; If there is a low complement and/or anti dsDNA antibody score, the clinical symptom score for SLEDAI-2000 (excluding low complement and/or anti dsDNA antibodies) must be ≥ 6 points;
* At least 6 months of stable standard treatment have been used in the SLE history prior to screening, and the condition remains active for at least 2 months prior to screening. The standard treatment plan refers to the stable use of any of the following drugs (used alone or in combination): glucocorticoids (≤ 20mg/day prednisone or equivalent), antimalarials (hydroxychloroquine ≤ 400mg/day, chloroquine ≤ 500mg/day), nonsteroidal anti-inflammatory drugs (NSAIDs), biologics (rituximab, belimumab, tacept), and other immunosuppressants or immunomodulators, including mycophenolate mofetil (≤ 2g/day), azathioprine (≤ 2mg/kg/day), methotrexate (≤ 20mg/week), etc;
* Recurrent/refractory dcSSc subjects must meet the following criteria:
* According to the 2013 EULAR/ACR classification criteria for systemic sclerosis (SSc), the diagnosis is SSc;
* According to the definition criteria of LeRoy et al. in 1988, it meets the diffuse skin type presentation, which refers to extensive skin fibrosis and involvement of the skin near the elbow and/or knee;
* When screening, interstitial lung disease (ILD) should be included, and 45% of the predicted values should be ≤ forced vital capacity (FVC) ≤ 70% of the predicted values, or 40% of the predicted values should be ≤ diffusion capacity of carbon monoxide (DLCO) ≤ 70% of the predicted values;
* Relapse/refractory is defined as: recurrence after previous ineffective conventional treatment or disease remission. Conventional treatment refers to the use of glucocorticoids, cyclophosphamide, and at least one immunosuppressive/regulatory drug for at least 6 months. Immunosuppressive/regulatory drugs include azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, rituximab, belimumab, tacrolizumab, etc;
* Activity is defined as having at least one of the following:

There is evidence of skin progression during screening, that is, an increase of ≥ 10% in mRSS scores within the past 6 months;

During screening, there is evidence of any of the following ILD activities:

Newly diagnosed ILD within the past 6 months; Previous ILD subjects had a 10% decrease in FVC or a 5% decrease in FVC accompanied by a 15% decrease in DLCO within the past 6 months.

* Recurrent/refractory AAV subjects must meet the following criteria:
* According to the definition of the 2012 Chapel Hill Consensus Conference (CHCC), clinical diagnosis is granulomatous vasculitis (GPA) and microscopic polyangitis (MPA);
* In Birmingham Vasculitis Activity Score (BVAS) version 3, at least one primary item or at least three other items;
* During screening, antibodies against PR3-ANCA or MPO-ANCA were positive;
* The definition of recurrence/refractory is:

Recurrent AAV subjects: those who have received initial efficacy (BVAS score 0 and glucocorticoid dose ≤ 7.5mg/d prednisone or other equivalent glucocorticoid drugs) after at least 3 months of combined glucocorticoid and immunosuppressive therapy (cyclophosphamide, rituximab, azathioprine, methotrexate, mycophenolate mofetil, etc.), and have experienced at least 1 disease recurrence (recurrence defined as the appearance of at least one important item in BVAS assessment, or at least 3 other items, or 1-2 new items in two consecutive assessments), and have experienced disease recurrence within 12 weeks before screening; Difficult to treat AAV subjects: Despite at least 3 months of previous treatment with corticosteroids combined with immunosuppressants (cyclophosphamide, rituximab, azathioprine, methotrexate, mycophenolate mofetil, etc.), no therapeutic effect has been achieved (BVAS score 0 and glucocorticoid dose ≤ 7.5mg/d prednisone or other equivalent glucocorticoid drugs);

* Recurrent/refractory IIM subjects must meet the following criteria:
* According to the 2017 EULAR/ACR IIM classification criteria, the probability of being diagnosed with IIM is ≥ 55%, and based on factors such as age of first onset, skin and muscle strength, laboratory tests, and muscle biopsy characteristics, it is classified as dermatomyositis (DM), polymyositis (PM), or immune-mediated necrotizing myopathy (IMNM):
* Disease activity/severity meets the following criteria:

Manual muscle strength check-8 (MMT-8) score ≤ 141 (total score of 150):

Meet at least 2 of the anomalies in other CSMs:

The overall disease activity evaluated by the patient [based on Visual Analog Scale (VAS)] score is ≥ 2 points (range 0-10 points); The overall disease activity VAS score evaluated by physicians is ≥ 2 points (range 0-10 points); The overall extramuscular disease activity VAS score evaluated by the physician is ≥ 2 points (range 0-10 points); The Health Assessment Questionnaire Disability Index (HAQ-DI) score evaluated by physicians is ≥ 0.25 (range 0-3 points).

At least one muscle enzyme level is greater than 1.5 times the upper limit of normal (ULN).

* Recurrent/refractory SS subjects must meet the following criteria:
* According to the 2016 EULAR/ACR SS classification criteria, the diagnosis is SS;
* Positive for anti Ro/SSA antibodies during screening;
* Dynamic saliva total flow rate ≥ 0.05 mL/min or static saliva total flow rate ≥ 0.01 mL/min during screening;
* Activity is defined as a Dry Syndrome Disease Activity Index (ESSDAI) score of ≥ 5 across 8 sub items;
* For autoimmune diseases that are intolerant to or have insufficient efficacy in the treatment of glucocorticoids and at least one other immunosuppressant or modulator in the past, it is required to be treated with glucocorticoids and at least two immunosuppressants (azathioprine, methotrexate, mycophenolate mofetil, etc.) at known effective doses for at least 3 months;
* Having good organ function:
* Blood routine: Absolute neutrophil count (ANC) ≥ 0.5 × 109/L, platelet count (PLT) ≥ 20 × 109/L, hemoglobin ≥ 60 g/L;
* Coagulation function: International normalized ratio (INR) ≤ 1.5 times ULN, and activated partial thromboplastin time (APTT) ≤ 1.5 times ULN;
* Liver function: serum aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 3 times the upper limit of normal (ULN), total bilirubin ≤ 1.5 times ULN;
* Renal function: serum creatinine ≤ 1.5 × ULN or creatinine clearance rate (Cockcroft Gault formula) ≥ 30 mL/min;
* Cardiac function: NYHA grade I or II, with an echocardiogram (ECHO) left ventricular ejection fraction (LVEF) ≥ 50% and no pericardial effusion; There were no clinically significant abnormal findings in the 12 lead electrocardiogram (ECG);
* Pulmonary function: Under indoor ventilation conditions, the oxygen saturation in non oxygenated state is ≥ 92%; No clinically significant pleural effusion;
* Expected survival period greater than 6 months;
* Subjects with reproductive partners agree to use effective contraceptive measures throughout the entire treatment period and for 24 months after treatment, and are not allowed to donate eggs/sperm for assisted reproduction during this period; Female subjects of childbearing age (those who have undergone sterilization surgery or have been menopausal for ≥ 12 months are not considered fertile) with negative urine pregnancy or blood pregnancy tests during the screening period; Voluntarily participate in this experiment and sign the informed consent form.

Exclusion Criteria:

* Subjects who meet any of the following criteria are not eligible for inclusion in this study:
* Patients with previous or concurrent active malignant tumors, including tumor associated polymyositis/dermatomyositis. Cervical carcinoma in situ that has been cured or has not recurred for at least 2 years, non-invasive basal cell or squamous cell skin cancer, locally treated prostate cancer, and ductal carcinoma in situ after radical surgery are excluded;
* Within the past 3 months, severe pulmonary diseases such as moderate to severe pulmonary arterial hypertension (average pulmonary arterial pressure detected by echocardiography>60 mmHg) require oxygen mask therapy or non-invasive or invasive ventilator assisted breathing during screening; During screening, IgA, IgG, and IgM levels were below the lower limit of normal (LLN);
* Patients who have used any of the following medications or treatments within the specified time:
* Individuals who have used B-cell depletion therapy within the previous month and have not failed treatment as assessed by clinical physicians, including those targeting CD20, CD22, CD52, CD38, BCMA monoclonal antibodies, or bispecific antibodies;
* Screening for excessive use of human intravenous immunoglobulin within the previous month;
* Use therapeutic doses of corticosteroids (prednisone ≥ 20mg/day or equivalent doses of other corticosteroids) within 24 hours prior to Qinglin pretreatment;
* Received corticosteroid shock therapy within 2 weeks (defined as a dose ≥ 500mg/d of prednisone or equivalent dose of other corticosteroids);
* Received tacrolizumab within 2 weeks prior to screening, or received belimumab within 3 weeks;
* Patients with a history of severe central nervous system diseases or related symptoms (excluding simple trigeminal nerve disease) within the past 6 months, including but not limited to: lupus encephalopathy, cerebrovascular disease, encephalitis, brain injury, aneurysm, cerebellar disease, organic brain syndrome, Parkinson's disease and other central nervous system diseases, as well as epilepsy, seizures, aphasia, dementia and other symptoms;
* Individuals who have experienced lupus crisis within the previous 3 months, such as active central nervous system lupus, severe hemolytic anemia, severe thrombocytopenic purpura, severe neutropenia, severe myocardial injury, severe lupus pneumonia or pulmonary hemorrhage, severe lupus hepatitis, severe vasculitis, etc;
* Concurrent severe kidney disease: severe lupus nephritis (defined as urinary protein>4g/24 hours or serum creatinine>1.5 × ULN or creatinine clearance rate (Cockcroft Gault formula)<30 mL/min) within the first 8 weeks of screening, Or active nephritis that requires treatment with drugs prohibited by the protocol, or requires treatment with prednisone greater than 500mg/day or equivalent corticosteroids for ≥ 14 days;
* Those who have severe allergies to the Qinglin pre-treatment drugs and any components of autologous CD19 CAR-T used in this study;
* hepatitis B surface antigen (HBsAg) positive and peripheral blood HBV DNA positive; Individuals with positive hepatitis C virus (HCV) antibodies and positive HCV RNA; Positive for Treponema pallidum antibody; HIV antibody positive individuals;
* There are uncontrolled fungi, bacteria, viruses, or other infections that researchers have assessed as unsuitable for participation in the study;
* History of major organ transplantation (such as heart and lung); During screening, there is active tuberculosis or latent tuberculosis (referring to whether the tuberculin skin test or interferon test is positive, and there are no clinical symptoms or imaging evidence);
* If any of the following cardiovascular diseases (including but not limited to) have occurred within the 6 months prior to screening:
* Congestive heart failure, myocardial infarction, unstable angina, coronary angioplasty, stent implantation, coronary artery/peripheral artery bypass grafting;
* Serious arrhythmias that require treatment (such as persistent ventricular tachycardia, ventricular fibrillation, apical torsion ventricular tachycardia, etc.); Congenital long QT syndrome, left anterior half block (double bundle block), allowing asymptomatic right bundle branch block to be included in the study;
* Uncontrolled hypertension (systolic blood pressure greater than 160 mmHg and/or diastolic blood pressure greater than 100 mmHg), history of hypertensive crisis or hypertensive encephalopathy;
* In addition to the target indication, patients with a history of other autoimmune diseases (including but not limited to eosinophilic granulomatous polyangitis, cryoglobulinemia vasculitis, inclusion body myositis, anti glomerular basement membrane disease, Behcet's disease or Takayasu arteritis, etc.) who require systematic treatment;
* Individuals with a family history of non IIM such as drug-induced myopathy or human immunodeficiency virus related myopathy;
* Pregnant or lactating women;
* Those who have received a live vaccine within 6 weeks before the pre-treatment of Qinglin;
* Participants who have participated in other interventional clinical studies, received active investigational drug treatment, or intended to participate in another clinical trial or receive treatment for autoimmune diseases outside of the protocol within 3 months prior to signing the informed consent form during the entire study period;
* Mental illness patients with depression or suicidal tendencies; The researchers believe that there are other factors that are not suitable for inclusion or affect the participation or completion of the study by the subjects.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 0~28 day after treatment

CONTACTS AND LOCATIONS:
Overall Officials: yajing zhang, MD/PhD, Principal Investigator — Beijing Gaobo Boren Hospital
Locations (1):
- Beijing Gobroad Brond Hospital, Beijing, Beijing Municipality, China